CLINICAL TRIAL: NCT02551133
Title: Comparison of the Two Different Doses of Dexamethasone on Persistent Mastectomy Pain
Brief Title: Comparison of Dexamethasone Doses on Persistent Postmastectomy Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Onur Koyuncu, Assist.Prof, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 208
Record Dates: First submitted 2015-09-07; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Mastectomy, Modified Radical
Keywords: Dexamethasone; mastectomy; persistent surgical pain
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.1 mg/kg dexamethasone (Active Comparator): 0.1 mg/kg dexamethasone intravenous will be given 1 h before surgery.
  Interventions: Drug: dexamethasone
- 0.2 mg/kg dexamethasone (Active Comparator): 0.2 mg/kg dexamethasone intravenous will be given 1 h before surgery.
  Interventions: Drug: dexamethasone

INTERVENTIONS:
Drug: dexamethasone — 1 hour before surgery

SUMMARY:
This study evaluates the effect of dexamethasone on persistent surgical pain after mastectomy operations. Half of the participants will receive 0.1 mg/kg dexamethasone and the other half will receive 0.2 mg/kg dexamethasone.

DETAILED DESCRIPTION:
Breast cancer is the most frequent malignancy of middle age women (%32) and causes 19% of cancer-related deaths. Acute pain can contribute to the development of persistent surgical pain. Persistent postsurgical pain has been demonstrated to be clinically relevant in 10% to 50% of patients undergoing various common operations, including breast cancer surgery. The pathogenic mechanisms are multiple, including nerve damage related to surgical technique resulting in risk of intercostobrachial neuralgia, neuroma pain, or phantom breast pain. Multimodal analgesic strategies are important.Glucocorticoid steroids can also provide beneficial effects when administered in appropriate doses as part of a multimodal analgesic regimen in the perioperative setting. A recent study demonstrated that preoperative application of dexamethasone reduced postoperative nausea and vomiting and pain in patients after thyroidectomy.. It is possible that the already established reduction in prostaglandin synthesis mediated by dexamethasone contributes to the analgesia. And also there are a lot of mechanisms more.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old, female patients
* Written informed consent.

Exclusion Criteria:

* American Society of Anesthesiologists Physical Status ˂3
* Any contraindication to dexamethasone
* Emergency or urgent procedure
* Obesity body mass index ≥27 kg m2
* Motion sickness and vertigo patients
* Axis I psychiatric disease (major depressive disorder, bipolar disorder, schizophrenia, etc.)
* Significant hepatic (Alanine aminotransferase or Aspartate aminotrans > 2 times normal)
* Renal (serum creatinine > 2 mg/dl) impairment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Persistent Surgical Pain on visual analogue scale (VAS). | Postoperative 3 months
  At 3.month persistent surgical pain will be evaluated using (visual analogue scale=VAS) (score ranges from O (no pain) to 10 (worst possible pain) . The difference between these VAS scores will be evaluated statistically.

SECONDARY OUTCOMES:
Change From Baseline in Acute Postsurgical Pain on visual analogue scale (VAS). | Postoperative 24 hours
  0.h, 1.h, 2.h, 4.h, 8.h, 12.h, 24.h (visual analogue scale=VAS) (score ranges from O (no pain) to 10 (worst possible pain) postoperative pain will be evaluated in the acute 24 h postoperative period

OTHER OUTCOMES:
Treatment-Related Adverse Events | Postoperative 24 hours
  For postoperative 24 hours (0.h, 1.h, 2.h, 4.h, 8.h, 12.h, 24.h) adverse events (Bradycardia, hypertension, headache, respirator depression, cough, bronchospasm) will be evaluated. At the end of this, all of the adverse events will be assessed statistically.

CONTACTS AND LOCATIONS:
Overall Officials: Onur Koyuncu, Assist.Prof, Principal Investigator — Mustafa Kemal University

REFERENCES:
- [Background] Worni M, Schudel HH, Seifert E, Inglin R, Hagemann M, Vorburger SA, Candinas D. Randomized controlled trial on single dose steroid before thyroidectomy for benign disease to improve postoperative nausea, pain, and vocal function. Ann Surg. 2008 Dec;248(6):1060-6. doi: 10.1097/SLA.0b013e31818c709a. PMID 19092351
- [Background] Vilholm OJ, Cold S, Rasmussen L, Sindrup SH. The postmastectomy pain syndrome: an epidemiological study on the prevalence of chronic pain after surgery for breast cancer. Br J Cancer. 2008 Aug 19;99(4):604-10. doi: 10.1038/sj.bjc.6604534. PMID 18682712